CLINICAL TRIAL: NCT05266872
Title: Biomaterial Collection for Neurodegenerative Disease Research (ND Collection)
Brief Title: Earlier Diagnosis and Better Treatment Mission Related to the Cohort Programme
Acronym: LuxPARK
Status: Recruiting | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: University of Luxembourg (Other); Laboratoire National de Santé (LNS) (Unknown); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: CNER 140174_ND
Record Dates: First submitted 2021-06-17; First posted 2022-03-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; longitudinal cohort; stratification; risk factors
MeSH Terms: conditions — Parkinson Disease | interventions — Observation; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At inclusion and Follow-up:
  Blood; Urine; Saliva
  Optional:
  Hair; Nasal washes; Nasal brushes; skin biopsy; Stool sample; Cerebrospinal Fluid Sample - lumbar puncture; Colorectal tissue sample (if colonoscopy required in SoC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD patients: Subjects with neurodegenerative disease or having degenerative parkinsonism (typical PD or atypical parkinsonism)
  Interventions: Other: Observational study with sample and data collection
- Healthy controls: Gender- and age-matched healthy controls
  Interventions: Other: Observational study with sample and data collection

INTERVENTIONS:
Other: Observational study with sample and data collection — Observational study with sample and data collection

SUMMARY:
The Luxembourg Parkinson's Study is an ongoing longitudinal nationwide monocentric observational study. It collects extensive clinical, molecular, genetic, and digital device-based longitudinal data, as well as foreseen post-mortem diagnostic validation (Hipp et al., 2018). The cohort consists of more than 1,600 participants from Luxembourg and the Greater Region, comprising patients with typical PD or atypical parkinsonism - irrespective of disease stage, age, cognitive status, comorbidities, or linguistic background - followed-up annually and age- and sex-matched healthy control subjects followed-up every 4 years. To provide a large, longitudinally followed, and deeply phenotyped set of patients and controls for clinical and fundamental research on PD, the investigators have implemented an open-source digital platform that has been partly harmonized with other international PD cohort studies. This effort is flanked by comprehensive biosampling efforts assuring high quality and sustained availability of body liquids and tissue biopsies (including blood, urine, stool, saliva, hair, skin biopsy and cerebrospinal fluid). All data and samples are stored, curated, and integrated into state-of-the-art data and biobank facilities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with neurodegenerative disease or having Parkinson's disease (typical PD or atypical parkinsonism)
* Subjects of all genders with a full capacity of consent
* Subjects with a limited consent capacity if the legal guardian/authorised representative is in agreement
* Subjects of at least 18 years of age at the time of inclusion

Exclusion Criteria:

* Refusal to sign the informed consent
* Limited capacity of consent on the part of the donor, if there is no legally determined guardian/authorised representative, or the latter is not present or does not agree with the inclusion
* Active cancer
* Pregnant women
* Underage subjects of less than 18 years of age
* Refusal to comply with mandatory sample collection
* For invasive procedures, i.e., lumbar puncture and skin biopsy: relevant blood clotting impairment, e.g., anamnestic evidence of frequent or prolonged bleedings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a neurodegenerative disease or having degenerative parkinsonism (typical PD or atypical parkinsonism) and gender- and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2014-12-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Establish an open collection of a large set of diverse longitudinal bio-samples and data for research in 800 PD patients and 800 controls | through study completion, an average of 8 years
  1.1. Samples will be aliquoted and stored according to the highest standards at the IBBL for future research.
2. Stratification of parkinsonism into subtypes and definition of individual progression trajectories of PD. | through study completion, an average of 8 years
  2.1. Identify PD patients' subgroups with a similar pattern of disease progression. datasets.
Determine Parkinson's disease biomarker signatures | through study completion, an average of 8 years
  3.1. Identify new and early diagnostic biomarkers
Develop a mechanistic understanding of the disease | through study completion, an average of 8 years
  4.1. Understand the mechanisms of PD pathogenesis.

SECONDARY OUTCOMES:
Inform future studies testing new therapies for Parkinson's disease | through study completion, an average of 8 years
  1.1. Enable future studies, such as clinical trials, by sharing the findings of mechanisms of PD pathogenesis and identifying new therapeutic targets.
Harmonization of data with international Parkinson's disease cohort studies | through study completion, an average of 8 years
  2.1. Data collected in this study will be harmonized with the international PD research community through an open-source digital platform.

CONTACTS AND LOCATIONS:
Overall Officials: Rejko Rejko, Dr, Principal Investigator — Luxembourg Institute of Health
Locations (2):
- Luxembourg (2):
  - Centre Hospitalier de Luxembourg (CHL), "Parkinson's Research Clinic", Luxembourg
  - Clinical and Epidemiological Investigation Center (CIEC), Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavelka L, Rawal R, Ghosh S, Pauly C, Pauly L, Hanff AM, Kolber PL, Jonsdottir SR, Mcintyre D, Azaiz K, Thiry E, Vilasboas L, Soboleva E, Giraitis M, Tsurkalenko O, Sapienza S, Diederich N, Klucken J, Glaab E, Aguayo GA, Jubal ER, Perquin M, Vaillant M, May P, Gantenbein M, Satagopam VP, Kruger R; NCER-PD Consortium. Luxembourg Parkinson's study -comprehensive baseline analysis of Parkinson's disease and atypical parkinsonism. Front Neurol. 2023 Dec 19;14:1330321. doi: 10.3389/fneur.2023.1330321. eCollection 2023. PMID 38174101
- See also: Website accessible by participants and researcher giving information on the study an related activities — https://parkinson.lu/
- See also: Publication on the initial cohort — https://www.frontiersin.org/articles/10.3389/fnagi.2018.00326/full